CLINICAL TRIAL: NCT01553786
Title: STUDY OF THE EFFICACY AND SAFETY OF FIRST LINE TREATMENT WITH CHOP AND LENALIDOMIDE (Rev-CHOP) IN PATIENTS AGED FROM 60 TO 80 YEARS WITH PREVIOUSLY UNTREATED ANGIOIMMUNOBLASTIC T-CELL LYMPHOMA (AITL)
Brief Title: Efficacy of a Treatment With CHOP and Lenalidomide in First Line in Angioimmunoblastic T-cell Lymphoma (AITL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REVAIL
Record Dates: First submitted 2012-01-20; First posted 2012-03-14 (Estimated); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: T-cell Lymphoma
Keywords: T-cell lymphoma; CHOp; lenalidomide
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lenalidomide (Experimental): lenalidomide + CHOP
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide

SUMMARY:
This study aims to evaluate the efficacy of lenalidomide associated with CHOP as measured by complete response rate at the end of treatment. Approximately 80 patients aged between 60 and 80 years will be included, to have 70 evaluable patients. The treatment consists of two phases of four 3-weeks cycles: induction phase and consolidation phase, for a total treatment duration of 24 weeks. Each cycle will be broken down as follows: chemotherapy will be administered in the hospital on day 1, prednisone is continued for 5 days and lenalidomide is taken for 14 days. Patients will be followed for at least 18 months after inclusion of the last patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven T-cell angioimmunoblastic lymphoma (AITL)
* Age from 60 to 80 years.
* Eastern Cooperative Oncology Group performance status 0 to 2.
* No previous therapy (except corticosteroids providing they have been initiated less than 15 days before inclusion).
* Spontaneous life expectancy > 1 month.
* Written informed consent. The Lenalidomide Information Sheet (in appendix N of the protocol) will be given to each patient receiving lenalidomide study therapy. The patient must read this document prior to starting lenalidomide study treatment and each time they receive a new supply of study drug.
* Male patients must:

  * Agree to use a condom during sexual contact with a FCBP, even if they have had a vasectomy, throughout study drug therapy, during any dose interruption and after cessation of study therapy.
  * Agree to not give semen or sperm during study drug therapy and for a period after end of study drug therapy.
* All patients must:

  * Have an understanding that the study drug could have a potential teratogenicity.
  * Agree to abstain from donating blood while taking study drug therapy and following discontinuation of study drug therapy.
  * Agree not to share study medication with another person.
  * Be counselled about pregnancy precautions and risks of foetal exposure.

Exclusion Criteria:

* Others categories of T-cell lymphoma.
* Central nervous system involvement by lymphoma.
* Any previous therapy for lymphoma except short-term corticosteroids (maximum 10 days) before inclusion.
* Contra-indication to any drug included in the CHOP regimen.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study (according to the investigator's decision).
* Active bacterial, viral or fungal infection, in particular active hepatitis B or C and HIV positive serological test.
* Impaired renal function (Creatinine clearance <50 ml/min (as calculated by the Cockcroft-Gault formula)) or impaired liver function tests (total bilirubin level > 30 µmol/L, transaminases > 2.5 upper normal limits) unless they are related to the lymphoma.
* Poor bone marrow reserve as defined by neutrophils < 1.0 x 109/L or platelets < 100 x 109/L, unless related to bone marrow infiltration.
* Any history of malignancy, other than that treated in this research, unless the patient has remained free of the disease for over 5 years.
* Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study.
* Hypersensitivity to the active substance or to any of the excipients.
* Pregnant and lactating woman
* Females of Childbearing potential (FCBP*) according to the Pregnancy Prevention Plan in appendix L of the protocol)

  * The Pregnancy Prevention Plan defines a female of childbearing potential as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Complete response rate | maximum 60 days after last study drug intake

CONTACTS AND LOCATIONS:
Overall Officials: Corinne HAIOUN, Principal Investigator — Lymphoma Study Association
Locations (30):
- Belgium (3):
  - Université Catholique de Louvain Saint Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Université Catholique de Louvain Mont Godinne, Yvoir
- France (27):
  - CHU d'Amiens - Hôpital Sud, Amiens
  - CHU Angers, Angers
  - CH d'Avignon - Hôpital Henri Duffaut, Avignon
  - CHU Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre hospitalier Chalon sur Saone William Morey, Châlon Sur Saône
  - CHU Estaing, Clermont-Ferrand
  - CH Sud Francilien de Corbeil, Corbeil-Essonnes
  - Hôpital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CH Départemental, La Roche-sur-Yon
  - CHRU de Lille, Lille
  - Institut Paoli Calmette, Marseille
  - Centre Hospitalier de Meaux, Meaux
  - CHU Saint-Eloi, Montpellier
  - CHU Hôtel Dieu, Nantes
  - Hôpital Saint Louis, Paris
  - Hôpital Necker, Paris
  - Centre Francois Magendie, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - Centre Hospitalier de la Région d'Annecy, Pringy
  - CHU Robert Debré, Reims
  - CHU Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - CHU Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lemonnier F, Safar V, Beldi-Ferchiou A, Cottereau AS, Bachy E, Cartron G, Fataccioli V, Pelletier L, Robe C, Letourneau A, Missiaglia E, Fourati S, Moles-Moreau MP, Delmer A, Bouabdallah R, Voillat L, Becker S, Bossard C, Parrens M, Casasnovas O, Cacheux V, Regny C, Camus V, Delfau-Larue MH, Meignan M, de Leval L, Gaulard P, Haioun C. Integrative analysis of a phase 2 trial combining lenalidomide with CHOP in angioimmunoblastic T-cell lymphoma. Blood Adv. 2021 Jan 26;5(2):539-548. doi: 10.1182/bloodadvances.2020003081. PMID 33496747